CLINICAL TRIAL: NCT03359720
Title: Knowledge Attitudes Behaviours and Practices Regarding HIV of Men Who Have Sex With Men in the French Antilles and French Guiana
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: INTERREG HSH
Record Dates: First submitted 2017-11-24; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- guyane
  Interventions: Other: no intervention survey
- martinique
  Interventions: Other: no intervention survey
- guadeloupe
  Interventions: Other: no intervention survey

INTERVENTIONS:
Other: no intervention survey — survey

SUMMARY:
determine the Knowledge attitudes behaviours and practices regarding HIV of men who have sex with men in the French Antilles and French Guiana

ELIGIBILITY:
Inclusion Criteria:

* men who have sex with men aged over 18

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — men who have sex with men
Study Population: men who have sex with men
Sampling Method: Non-Probability Sample
Enrollment: 766 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge attitudes behaviours and practices regarding HIV of men who have sex with men in the French Antilles and French Guiana - Questionnaire Survey | one year

IPD SHARING:
Plan to Share IPD: No